CLINICAL TRIAL: NCT02929615
Title: Study of Standard and Individualized Treatment Model for Relapse and Refractory Lymphatic System Malignant Tumors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v1.0-20150805
Record Dates: First submitted 2016-09-27; First posted 2016-10-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Hematopoietic Stem Cell Transplantation

ARMS (1):
- Treatment group (Experimental)
  Interventions: Other: Hematopoietic stem cell transplantation

INTERVENTIONS:
Other: Hematopoietic stem cell transplantation

SUMMARY:
The purpose of the study is to research the standard and individualized treatment model for relapse and refractory lymphatic system malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapse and refractory lymphoma and multiple myeloma.
2. At least 1 measurable lesions and its size≥15mm.
3. Patients ≤65 years，no limitations for both gender.
4. ECOG score is 0-1.
5. Life expectancy≥3 months.
6. LVEF≥ 55%; Peripheral blood: WBC ≥ 3.5×10(9)/L,neutrophil ≥1.5×10(9)/L, PLT≥75×109/L，Hb≥90g/L; Renal function: Cr≤2.0×UNL; Liver function: BIL≤2.0×UNL，ALT/AST≤2.5×UNL;
7. Written informed consent are acquired.

Exclusion Criteria:

1. Previously received stem cell transplantation.
2. Women with pregnant, lactating or not to take contraceptive measures.
3. Severe acute infection or suppurative and chronic infection that wound not healing.
4. Severe heart failure.
5. Suffering from mental disorders and poor compliance.
6. Other situations that investigators consider as contra-indication for this study.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 2 years after treatment
complete response | 2 years after treatment
progression-free survival | 2 years after treatment
overall survival | 2 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing Municipality, China